CLINICAL TRIAL: NCT07226401
Title: Preventing Intimate Partner Violence Among Teens Who Are Pregnant or Parenting
Brief Title: Virtual Village for Young Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Marni Kan, Senior Research Public Health Analyst 1, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD111729 (NIH); R21HD111729 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gender-based Violence; Intimate Partner Violence
Keywords: Young Adult Parents; Adolescent Pregnancy

STUDY DESIGN:
Intervention Model Description: Individual adolescent and young adults (AYA) will be block-randomized to the SDYP intervention (intervention condition) or an equal attention control condition using a 1:1 allocation to ensure balanced assignment, using permuted blocks sizes of 4 and 6. The field data collector will be blinded to the group assignment until after baseline data collection is completed. They will notify each participant of their assigned condition. Implementation staff (i.e. the facilitators) will also be informed about each participant's assignment so that they can support participation in the SDYP intervention for those randomized to the intervention condition or control implementation for those randomized to the control. Both intervention and control programs will be implemented with closed virtual groups of five or more participants; study staff will be responsible for scheduling groups and ensuring attendance. Sessions will be implemented separately from any other agency programs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Safe Dates for Young Parents (Experimental): Participants assigned to the intervention group will be offered the Safe Dates for Young Parents (SDYP) program activities focused on healthy relationships and intimate partner violence (IPV) prevention. This program will consist of 10 modules, with sessions that are 60-90 minutes each. The intervention will be done with groups via zoom and will be led by a trained facilitator.
  Interventions: Behavioral: Virtual Safe Dates for Young Parents
- HealthSmart (Active Comparator): The study will use an equal attention control condition where control group participants will be offered lessons on physical activity and nutrition from the HealthSmart digital high school curriculum. To achieve consistent dosage with SDYP, ten lessons will be chosen from the curriculum. This program will not provide education about IPV or healthy relationships content that composes the SDYP intervention. The intervention will be done with groups via zoom and will be led by a trained facilitator.
  Interventions: Behavioral: HealthSmart

INTERVENTIONS:
Behavioral: Virtual Safe Dates for Young Parents — Safe Dates for Young Parents (SDYP) is a healthy relationship and intimate partner violence (IPV) prevention program, adapted from "Safe Dates (Foshee et al., 1998; Foshee et al., 1996)" for pregnant or parenting young adults. The investigators adapted the prevention curriculum and related intervention materials for virtual delivery via Zoom. The program consists of ten group-based sessions (50 minutes of content each) led by a trained facilitator. The program includes interactive discussions, analysis of scenarios, games, role-plays, and brainstorming.
  Arms: Virtual Safe Dates for Young Parents
Behavioral: HealthSmart — The HealthSmart program will use 10 digital high school curriculum lessons focused on physical activity and nutrition. The sessions will be formatted appropriately to be delivered via zoom. Participants may be asked to complete handouts, listen to presentations, and participate in discussions. Topics may include information about different nutrients, how nutrients affect health, how to read food labels, healthy eating, and guidelines for physical activity.
  Arms: HealthSmart

SUMMARY:
This project will study virtual delivery of Safe Dates for Young Parents (SDYP), a 10-session, group-based intimate partner violence (IPV) prevention program tailored for adolescents and young adults who are pregnant or parenting. This program has the potential to improve the health and well-being of young parents and their children, and virtual delivery may improve participants' ability to attend. The main questions it aims to answer are: (1) Is it feasible and acceptable to implement SDYP in a virtual setting? (2) Are SDYP participants less likely to experience IPV than participants in an alternate health education program? Participants will be invited to a series of virtual program sessions for either SDYP or a health education program focused on physical activity and nutrition and will be asked to complete surveys before the programs begin and up to 6 months later.

DETAILED DESCRIPTION:
As many as two-thirds of teens who are pregnant or parenting have been the victims or perpetrators of physical intimate partner violence (IPV) and there is an even higher prevalence of psychological abuse in this population. IPV can endanger teen mothers' own health, the health of their pregnancies, and the well- being of their children. Despite this detrimental impact, there is a lack of evidence-based IPV prevention programs that are tailored for pregnant and parenting teens. Moreover, despite the promise of virtual program delivery, which may help improve teens' ability to attend, research has yet to determine feasibility and outcomes of virtual delivery of IPV prevention programs for teens who are pregnant or parenting. This study is a pilot test of the Safe Dates for Young Parents (SDYP) program adapted for virtual delivery. The original Safe Dates is a 10-session, theoretically based, interactive program with demonstrated efficacy in preventing psychological, physical, and sexual dating abuse among teens. The investigators previously adapted Safe Dates for young parents who are pregnant or parenting by integrating pregnancy and parenting themes throughout program sessions, increasing the focus on overcoming barriers to seeking help for intimate partner violence (IPV), and revising sexual assault content. The programs were delivered exclusively in person. A virtual approach to delivery could improve scale-up of SDYP, via increased reach and lower costs. The investigators recently pre-tested selections from the SDYP program over Zoom with 9 young parents to adapt the prevention curriculum and related intervention materials for virtual delivery. In this study, the investigators will build on this work by evaluating the virtual SDYP intervention in a pilot randomized trial to assess implementation outcomes (i.e. feasibility, acceptability, fidelity, and appropriateness) and preliminary effects on IPV outcomes. The study will randomize 80 individual pregnant and parenting young people 1:1 to intervention (SDYP) or equal attention control (virtual health education program lessons that do not address IPV) conditions, and conduct surveys at baseline and 3-6-month follow-up to assess IPV and related behavioral outcomes. The investigators will assess implementation outcomes (feasibility, acceptability, fidelity, and appropriateness) through program data, qualitative in-depth interviews (IDIs) with facilitators and participants, and survey data from the intervention group. Research activities will be done virtually with participants recruited from several locations around the United States.

ELIGIBILITY:
Inclusion Criteria:

Pregnant or parenting youth (Pilot RCT participants)

* Aged 16-21 years.
* Currently pregnant, partner of a pregnant person, or parenting a child (i.e., have contact with child at least once per week).
* Able to speak and read English.
* Willing and able to provide written informed consent.
* Willing and able to provide adequate contact/locator information.

Facilitators (IDI participants)

* Aged 18 years or older.
* Trained and served as a facilitator of the virtual SDYP intervention.
* Able to speak and read English.
* Able and willing to provide verbal informed consent.

Exclusion Criteria (Pilot RCT participants):

* Has any other condition that, in the opinion of the PI or their designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Currently participating or will be participating in a violence prevention education program in the next 3 months.
* Previously participated in the Empowering Young Parents study.

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Participant attendance | From the first to the last session of SDYP (typically 10 weeks)
  Percent of sessions attended (out of 10)
Participant engagement | From the first to the last session of SDYP (typically 10 weeks)
  Average of facilitator reports of participant engagement across SDYP sessions on a 4-point scale
Program adherence | From the first to the last session of SDYP (typically 10 weeks)
  Percent of SDYP activities completed without changes, averaged across sessions and facilitators
Physical IPV perpetration | Past 3 months measured at baseline and 3 to 6 months after baseline
  Endorsement of any of 7 items describing physically aggressive acts toward a partner, adapted from the WHO instrument and Safe Dates questionnaire measure
Physical IPV victimization | Past 3 months measured at baseline and 3 to 6 months after baseline
  Endorsement of any of 7 items describing physically aggressive acts by a partner, adapted from the WHO instrument and Safe Dates questionnaire measure
Psychological IPV perpetration | Past 3 months measured at baseline and 3 to 6 months after baseline
  Endorsement of any of 9 items describing psychologically aggressive acts toward a partner, adapted from the Safe Dates questionnaire measure
Psychological IPV victimization | Past 3 months measured at baseline and 3 to 6 months after baseline
  Endorsement of any of 9 items describing psychologically aggressive acts by a partner, adapted from the Safe Dates questionnaire measure

CONTACTS AND LOCATIONS:
Locations (1):
- RTI International, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Restricted access study data and associated documentation will be made available to the research community free of charge through a self-publishing repository for social, behavioral, and health sciences research data. Participants' identifying information (names and contact information) will not be included in shared data.
Time Frame: Submission of the study data will occur by the end of the project period.
Access Criteria: Restricted access study data and associated documentation will be made available to the research community free of charge through openICPSR. Given the sensitive nature of the teen survey data and the small sample sizes in the interview data, it is expected that these data will be designated as restricted-use data. ICPSR requires an application to access such data. As part of the application process, the data user must enter into a Restricted Data Use Agreement with ICPSR among other application components and data security requirements.